CLINICAL TRIAL: NCT00638196
Title: Phase II Study of Linoleic Acid in Relapsing Multiple Sclerosis
Brief Title: Placebo vs. Linoleic Acid Controlled Assessment of Treatment Efficacy in MS
Acronym: PLACATE-MS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: funding stopped due to slow enrollment.
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Andrew Goodman, MD, University of Rochester
Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 22084
Record Dates: First submitted 2008-03-10; First posted 2008-03-18 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Multiple Sclerosis
Keywords: relapsing multiple sclerosis; polyunsaturated fatty acids; omega-6 fatty acids
MeSH Terms: conditions — Multiple Sclerosis | interventions — Sunflower Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): placebo/active crossover
  Interventions: Drug: Linoleic Acid/Oleic Acid

INTERVENTIONS:
Drug: Linoleic Acid/Oleic Acid — Dietary Supplement: Linoleic acid emulsion 30g bid/Oleic acid emulsion 30g bid
  Other Names: sunflower oil

SUMMARY:
Several investigations have suggested that polyunsaturated fatty acids may promote therapeutic effects in MS. This pilot study will determine whether omega-6 polyunsaturated fatty acids (PUFAs),in the form of linoleic acid,can reduce disease activity and prevent disability progression in patients with relapsing MS.This study will seek to measure disease activity as seen on MRI scans in addition to measuring relapse rates.

DETAILED DESCRIPTION:
Participants who meet inclusion criteria will start placebo treatment by taking olive oil for 2 months. This period will include screening activities including 3 monthly MRIs. Those with 2 enhancing lesions on three placebo run-in period MRIs will continue in the study and receive omega-6 PUFA (linoleic acid) for 6 months. Brain MRIs will be repeated after 4,5, and 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsing MS
2. treated with FDA-approved dosage of interferon-beta (Avonex,Betaseron,Rebif), glatiramer acetate for at least 6 months OR no immunotherapy for at least 3 months
3. at least one clinical exacerbation or at least one gadolinium enhancing lesion on brain MRI in the past 12 months
4. at least two gadolinium enhancing lesions on three brain MRIs obtained during the placebo run-in period
5. women of childbearing potential may participate provided that they are using adequate birth control methods for the duration of the study. Women of childbearing potential must have a negative pregnancy test at baseline and be non-lactating.
6. willing and able to provide informed consent

Exclusion Criteria:

1. corticosteroids within 1 month prior to screening
2. treatment with other immunotherapies (other than interferon-beta, glatiramer acetate or sporadic corticosteroids) within 3 months prior to screening
3. any significant medical condition or laboratory abnormality which may interfere with the subject's ability to participate in the study, including peptic ulcer disease, avascular necrosis and hepatic insufficiency
4. history of hypersensitivity or intolerability to vegetable oils or their constituents
5. unable to perform any of the required study procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Within patient change in the sum of gadolinium-enhancing lesions on brain MRIs obtained during the treatment period compared to pre-treatment. | 9 months

SECONDARY OUTCOMES:
Annualized relapse rate | 9 months
Changes in depression and fatigue symptoms on standardized questionnaires (Beck Depression Scale and Modified Fatigue Impact Scale). | 9 months
Changes in T2 lesion counts/volume, change in T1 hypointense lesion counts/volume, white matter volume and gray matter volume | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Goodman, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States